CLINICAL TRIAL: NCT05318807
Title: A Personalised Prehabilitation Model for Patients Undergoing Chemotherapy, Radiotherapy and/or Immunotherapy Treatment for Lung Cancer: A Feasibility Pilot Study
Brief Title: Personalised Diet, Exercise and Emotional Support for Lung Cancer Patients Having Chemotherapy, Radiotherapy or Immunotherapy Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22CX7570
Record Dates: First submitted 2022-03-15; First posted 2022-04-08 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
Keywords: prehabilitation; radiotherapy; chemotherapy; feasibility; immunotherapy; nutrition; physical activity; psychological wellbeing
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Health Services Needs and Demand

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalised prehabilitation (Experimental): A personalised plan of diet, exercise and emotional support for patients having chemotherapy, radiotherapy and/or immunotherapy treatment for lung cancer.
  Interventions: Other: Assessment of level of readiness and need for personalised prehabilitation; Other: Formation of a personalised prehabilitation plan; Other: Daily diary

INTERVENTIONS:
Other: Assessment of level of readiness and need for personalised prehabilitation — Patients asked to complete five validated questionnaires to assess their level of need and readiness:
  1. Cancer Behaviour Inventory brief form - to measure self-efficacy for coping with cancer
  2. Patient Activation Measure - to measure patient activation
  3. Modified Godin Leisure Time Exercise Questionnaire - to monitor activity
  4. Patient Generated Subjective Global Assessment - to identify malnutrition risk
  5. Emotions thermometer - to detect emotional disorders and identify risk
Other: Formation of a personalised prehabilitation plan — Prior to starting treatment, at week three and at week six, each patient will be invited to see a specialist dietitian for a one hour face-to-face personalised prehabilitation appointment to:
  * Review the initial questionnaires to inform the personalised plan and goal setting
  * Complete a further four questionnaires related to quality of life, diet and exercise
  * Measure handgrip strength
  * Assess functional capacity by completing the six minute walk test
  A personalised plan is then agreed using SMART goals, taking into account the patient's priorities as indicated in their Patient Generated Index.
Other: Daily diary — Each patient will be asked to keep a daily diary to record their symptoms, appetite, mobility and mood throughout their treatment as well as their adherence to goals. This will provide an indication of the impact of symptoms.

SUMMARY:
Background

The term 'prehabilitation' refers to a period of time before treatment and often includes diet, exercise and/or wellbeing plans to help patients through their cancer treatment. Prehabilitation has shown to benefit patients having surgery, but there is little research into its use in the oncological setting.

The United Kingdom sees more deaths from lung cancer than any other cancer. 70-80% of lung cancer patients receive oncological treatment. Treatment side effects can have a significant impact on quality of life. Personalised prehabilitation can take into account the challenges patients face, helping patients through treatment.

Aim

To see if a personalised plan of diet, exercise and emotional support can be used in practice for patients having chemotherapy, radiotherapy and/or immunotherapy treatment for lung cancer.

Methods

The study will involve lung cancer patients from Imperial College Healthcare NHS Trust who are:

* Over the age of 18 years old
* Have not had previous lung cancer surgery and
* Are about to start chemotherapy, radiotherapy or immunotherapy treatment

The prehabilitation interventions will be based upon patient need and readiness, assessed using:

* A series of questionnaires
* An assessment of walking
* A measure of grip strength

These will be done prior to, at week three and at week six of a patient's oncological treatment regime. Personalised goals will be agreed at each stage.

Throughout treatment, patients will be asked to keep a daily diary to record their symptoms, appetite, mobility and mood. The diary will also be used to monitor goal adherence.

Public involvement

Patients will be part of a study advisory group, helping with research design and dissemination e.g. with the presentation of findings to the lung cancer support group.

Dissemination

All patients will receive a written summary of findings. Results will be shared in a scientific journal and presented at relevant conferences. Patients will not be identifiable.

DETAILED DESCRIPTION:
Background

Prehabilitation programmes are increasingly used before surgery to optimise outcomes. However, 55% of patients are treated non-surgically with oncological treatment. Prehabilitation has potential to increase resilience to withstand anticipated treatment deconditioning, but few prehabilitation pathways exist in the non-surgical field.

This is particularly the case for lung cancer, where 70-80% of patients have non-surgical treatment without access to prehabilitation. United Kingdom deaths from lung cancer are higher than any other cancer and outcomes are poor, highlighting an unmet need.

Study design

This is a study to assess if a personalised plan of diet, exercise and emotional support can be used in practice for patients having chemotherapy, radiotherapy and/or immunotherapy treatment for lung cancer.

To tackle the unmet need within the field of lung cancer, I have co-designed a personalised prehabilitation model with healthcare professionals and patients, informed by theory and evidence. It embodies personalised care with interventions stratified according to need and readiness. However, before I can trial it with lung cancer patients, there are key uncertainties that need to be resolved, including whether patients will sign up, engage and adhere to the prehabilitation interventions.

Methods

The study will involve lung cancer patients from Imperial College Healthcare National Health Service (NHS) Trust who are:

* Over the age of 18 years old
* Have not had previous lung cancer surgery and
* Are about to start chemotherapy or radiotherapy treatment

Patients will be identified by a member of their direct clinical care team, which will be either their lung consultant or their Clinical Nurse Specialist (CNS) from the weekly lung cancer meeting and a referral will be sent to the research team.

A sample size of 30 patients over a 6-month recruitment period is suitable within the time frame of this study and is based upon a recommend sample size of 24 - 50 for a pilot study.

Each patient will receive a patient information sheet either in person or electronically via email depending on their preference. If they agree to participate, they will be asked to complete a written consent form either in person or via email using their personal computer. Following consent, each patient will be asked to complete five validated questionnaires, either on paper or online. The five questionnaires will take approximately 30 minutes to complete. These five questionnaires will be used to assess a patient's level of readiness and need.

Each patient will then be invited to see a specialist dietitian for a separate one hour face-to-face personalised prehabilitation appointment at Charing Cross Hospital to:

* Review the initial questionnaires
* Complete a further four validated questionnaires related to quality of life, diet and activity (= 9 questionnaires in total)
* Measure grip strength. This will involve a patient sitting in a chair. The dietitian will ask the patient to squeeze the device as hard as they can using their non-dominant arm. Each patient will repeat this three times and the dietitian will record the average
* Undergo an assessment of walking. This will involve a patient walking at their own pace as far as they can in 6 minutes

The above assessments will then be repeated at week three and week six of a patients oncological treatment regime. Personalised goals will be agreed at each stage.

Owing to the nature of the above appointments and the need for measurements to be taken, a virtual consultation would not be practical.

Throughout treatment, patients will be asked to keep a daily diary to record their symptoms, appetite, mobility and mood. The diary will be given to patients by the research team at the start for the duration of the study. The research team will not need these to be sent back to them. Patients will receive a weekly telephone call to see how they are getting on. The language used during the phone calls and the face to face consultations is effective for building self-efficacy and to sustain behaviour change. Validation and compassion is at the core.

The personalised prehabilitation model is in line with the Macmillan universal, targeted and specialist approach for prehabilitation. All patients will receive universal interventions which involve signposting for support and/or information on emotional support, nutrition and/or exercise as required. If a patient identifies an emotional, nutritional and/or exercise need, they will then receive the appropriate intervention according to their level of need and readiness.

All patients who participate in the study will be offered the opportunity to provide feedback on their experience of the personalised prehabilitation model via the use of a short free text questionnaire. This feedback will be invaluable, as it will help inform future model adjustments and will have the potential to improve patient experience.

All patients will be given a unique study number that will be used from the start of the study. All data will be stored stored securely in accordance with the Trust policy on either a Trust computer, password protected, or under lock and key. Patient data will not be shared with parties outside of the patient's direct clinical care team or local research team.

The data will be analysed by the research team and all patients will receive a written summary of the findings. The results will be also be shared in scientific journals and conferences, so that others can learn from this as well. Patients will not be identifiable from any report or publication.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥ 18 years) diagnosed with lung cancer
* Able to give informed consent
* Due to embark on a chemotherapy, radiotherapy and/or immunotherapy treatment pathway

Exclusion Criteria:

* On a surgical pathway
* Have had previous lung cancer surgery
* Unable to understand verbal or written English
* Unable to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasible eligibility, recruitment and refusal rates | Immediately after week six of oncological treatment
  Use of descriptive statistics - number approached, eligible, recruited, refused
How many participants do not participate in the personalised prehabilitation programme and explore the reasons why | Immediately after week six of oncological treatment
  Use of descriptive statistics, field notes taken during the Lung Cancer Multi-Disciplinary Team (LCMDT) and participant discussion
Number of participants who are not suitable for the personalised prehabilitation programme and the reasons why | Immediately after week six of oncological treatment
  Use of descriptive statistics and field notes taken during the LCMDT, where discussions of eligibility will take place
Attrition rate throughout the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Use of descriptive statistics - number who drop out and at what stage
Number of participants who adhere to the goals set for the personalised prehabilitation interventions | Immediately after week six of oncological treatment
  Adherence to goals set measured through participant discussion at the weekly telephone consultations
Barriers and facilitators to adherence and intervention fidelity | Immediately after week six of oncological treatment
  Use of a daily diary - symptom log, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of the emotion thermometer questionnaire used for the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of the modified Godin leisure time exercise questionnaire used for the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of the patient generated subjective global assessment questionnaire used for the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of the patient activation measure questionnaire used for the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of the cancer behaviour inventory questionnaire used for the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of the patient generated index used for the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of measuring body weight in kilograms for the personalised prehabilitation progamme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of measuring functional capacity by the distance covered in meters using the six minute walk test as part of the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of participant acceptability of measuring grip strength in kilograms using a handgrip dynamometer as part of the personalised prehabilitation programme | Immediately after week six of oncological treatment
  Completion rates, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Evaluation of contextual or implementation factors which may influence acceptability of the intervention/s | Immediately after week six of oncological treatment
  Use of a daily diary - symptom log, discussions had with participants during the weekly telephone consultations; participant reflection, participant needs and priorities, short free text questionnaire at the end of the study, analysed thematically
Evaluation of contextual or implementation factors which may influence effectiveness of the intervention/s | Immediately after week six of oncological treatment
  Use of a daily diary - symptom log, discussions had with participants during the weekly telephone consultations; participant reflection, participant needs and priorities, short free text questionnaire at the end of the study, analysed thematically
The 'prehabilitation window' (length of time between diagnosis and the start of treatment) | Immediately after week six of oncological treatment
  Use of descriptive statistics - date of diagnosis, date of start of treatment, date of start and finish of prehabilitation
The extent to which the prehabilitation programme has had an impact on psychological wellbeing | Immediately after week six of oncological treatment
  Use of the emotional thermometer questionnaire which will be used to assess psychological wellbeing - change between baseline and follow up, daily diary - symptom log, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
The extent to which the prehabilitation programme has had an impact on nutrition | Immediately after week six of oncological treatment
  Use of the Patient Generated Subjective Global Assessment (PG-SGA) tool which will be used to assess nutritional status - change between baseline and follow up, daily diary - symptom log, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
The extent to which the prehabilitation programme has had an impact on physical activity | Immediately after week six of oncological treatment
  Use of the Modified Godin leisure time exercise questionnaire which will be used to assess physical activity - change between baseline and follow up, daily diary - symptom log, discussions had with participants during the weekly telephone consultations, short free text questionnaire at the end of the study, analysed thematically
Number of participants who require universal, targeted and specialist intervention | Immediately after week six of oncological treatment
  Use of questionnaires to assess level of need and readiness and descriptive statistics

SECONDARY OUTCOMES:
Quality of life assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQC30 questionnaire | Baseline; pre-treatment, during treatment and immediately after treatment
  Incidence of change between baseline and immediately after treatment assessed by any differences in the EORTC questionnaire
Quality of life assessed using the EuroQOL Group EQ-5D-5L questionnaire | Baseline; pre-treatment, during treatment and immediately after treatment
  Incidence of change between baseline and immediately after treatment assessed by any differences in the EQ-5D-5L questionnaire
Patient experience | Immediately after week six of oncological treatment
  Assessed via a short free text questionnaire. Patients will be able to openly give written feedback on their experience and offer any comments or suggestions
Functional capacity | Baseline; pre-treatment, during treatment and immediately after treatment
  Assessed by patients undertaking a six minute walk test
Handgrip strength | Baseline; pre-treatment, during treatment and immediately after treatment
  Assessed using a handgrip dynamometer to measure grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Wade-Mcbane, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All participants will be given a unique study number that will be used from the start of the study. Files (e.g. paper consent forms and questionnaires) will be stored in research offices and secured by either lock and key or key code and accessible by only departmental staff or the Trust's security department. Personal data (e.g. patient demographics and results of assessments) will be retained and stored on a networked and password protected NHS computer. Patient data will not be shared with parties outside of the patient's direct clinical care team or local research team.
  Stored data will be pseudonymised at the time of collection/storage. Data will be collected according to the data protection act 2018 and in line with general data Protection regulation GDPR).
  Results will be shared in a scientific journal and presented at relevant conferences. Patients will not be identifiable.

REFERENCES:
- [Derived] Wade-Mcbane K, King A, Urch C, Johansson L, Wells M. Is personalised prehabilitation feasible to implement for patients undergoing oncological treatment for lung cancer at a London teaching hospital? Protocol of a feasibility trial. BMJ Open. 2023 Jul 17;13(7):e072367. doi: 10.1136/bmjopen-2023-072367. PMID 37460263